CLINICAL TRIAL: NCT04592835
Title: A Double-blind, Randomized, Placebo-controlled, Single-ascending Dose Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetic Properties of Niclosamide Injectable (DWRX2003) Following Intramuscular Administration in Healthy Volunteers
Brief Title: To Evaluate the Safety, Tolerability and Pharmacokinetic Properties of DWRX2003
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWJ1516101_Australia
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: COVID-19 Patients

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (288mg) (Experimental): 72 mg/0.3 mL x 4 injection sites
  Interventions: Drug: DWRX2003
- Cohort 2 (576 mg) (Experimental): 144 mg/0.6 mL x 4 injection sites
  Interventions: Drug: DWRX2003
- Cohort 3 (960 mg) (Experimental): 216 mg/1.0 mL x 4 injection sites
  Interventions: Drug: DWRX2003

INTERVENTIONS:
Drug: DWRX2003 — Intramuscularly injection at predefined injection sites
  Drug: Placebo Intramuscularly injection at predefined injection sites

SUMMARY:
This study is designed to assess the safety, tolerability and Pharmacokinetic Properties of Niclosamide Injectable (DWRX2003) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, between 18 and 65 years of age, inclusive, at time of signing the Informed Consent Form (ICF).
2. Body mass index between 18.0 lesser than or equal to Body Mass Index (BMI) lesser than or equal to 32 at Screening, with a minimum weight of 50 kg (inclusive).
3. Willing to sign ICF on a voluntary basis and to voluntarily participate in the study, after being fully informed of and completely understanding this study, prior to any Screening procedure being undertaken

Exclusion Criteria:

1. Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the follow-up period;
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee). Please note participants with allergies which can be managed without treatment can be included based on the decision of the Investigator (or designee).
3. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-10-19 (Estimated); Primary Completion 2020-12-13 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | follow-up 35 days after dosing
  Incidence, severity and causality of adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
To assess PK parameters of niclosamide injectable (DWRX2003) through Cmax | at Day 1, 2, 3, 5, 7, 10, 14, 21 and 28
  Measured through Maximum (peak) plasma drug concentration (Cmax)
To assess PK parameters of niclosamide injectable (DWRX2003) through tmax | at Day 1, 2, 3, 5, 7, 10, 14, 21 and 28
  Time to reach Cmax following IP administration (tmax)
To assess PK parameters of niclosamide injectable (DWRX2003) through AUC0-last | at Day 1, 2, 3, 5, 7, 10, 14, 21 and 28
  Area under the curve from zero to time of last measurable concentration (AUC0-last)
To assess PK parameters of niclosamide injectable (DWRX2003) through AUC0-∞ | at Day 1, 2, 3, 5, 7, 10, 14, 21 and 28
  Area under the curve from zero to infinity (AUC0-∞)
To assess PK parameters of niclosamide injectable (DWRX2003) through t1/2 | at Day 1, 2, 3, 5, 7, 10, 14, 21 and 28
  Elimination half-life (t1/2)

IPD SHARING:
Plan to Share IPD: No